CLINICAL TRIAL: NCT03667586
Title: The Impact of Group Cognitive Behavioral Psychotherapy on Disease Severity and Psychosocial Functioning of Inflammatory Bowel Disease Patients
Brief Title: Group Cognitive Behavioral Therapy for IBD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Christos Triantos, Assistant Professor in Internal Medicine and Gastroenterology, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 326/15.05.2018
Record Dates: First submitted 2018-09-09; First posted 2018-09-12 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: The study design will be randomized prospective with a control group. More specifically, all patients will be randomly assigned either to the psychotherapy or the control group. Randomization will be 1:1 and will be performed through the method of sealed envelopes. A group of participants will receive weekly group cognitive behavioral therapy sessions, while another group will receive care as usual with regular weekly brief follow-ups by the gastroenterologists and the nurse of the research team. In total, the psychotherapeutic intervention will last for 6 months with participants attending weekly sessions for the first 3 months and monthly follow-up sessions for the next 3 months. All patients will be re-evaluated at 6 months (treatment completion), 12 months and 18 months after study initiation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Cognitive Behavioral Therapy (Experimental): Cognitive behavioral psychotherapy sessions will be conducted at an appropriately accommodated office of the Psychiatry Department in groups of 6-10 patients and will be coordinated by a qualified psychologist of the research team. Each session will be of 90 minutes duration. The initial two sessions will be psycho-educational and the remaining sessions will be based on the principles of Cognitive Behavioral Therapy (CBT). In total, the psychotherapeutic intervention will last for 6 months with participants attending weekly sessions for the first 3 months and monthly follow-up sessions for the next 3 months.
  Interventions: Behavioral: Group cognitive behavioral therapy
- Standard care (Placebo Comparator): Regular brief follow-ups by the gastroenterologists and the nurse of the research team
  Interventions: Behavioral: Group cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Group cognitive behavioral therapy — Group sessions based on the principles of Cognitive Behavioral Therapy and adjusted for chronic disease patients

SUMMARY:
Inflammatory bowel disease (IBD) patients commonly suffer from disturbed psychosocial functioning and poor quality of life compared to other chronic disease patients. Clinicians are becoming growingly aware that addressing patients' psychological difficulties may improve disease management, however, there is not adequate evidence regarding the effect of psychotherapeutic interventions on psychosocial functioning and disease-related clinical and laboratory parameters. The aim of the present study is the evaluation of the effects of a targeted, cognitive behavioral psychotherapeutic intervention on symptom severity, levels of psychological distress and quality of life and inflammation and disease activity indices in IBD patients. An additional aim is the detection of psychological and biomedical parameters which may be associated with these effects.

DETAILED DESCRIPTION:
Background Inflammatory bowel disease patients report increased levels of anxiety and depressive symptoms which are associated with poorer health-related quality of life (QoL). In addition, they commonly experience disturbed self- and body-image thus being vulnerable to interpersonal difficulties and sexual dysfunction. There are several studies reporting that the presence of co-morbid depression is more strongly associated with increased financial cost and hospitalization rates, worse treatment compliance and major QoL deficits compared to disease activity. For this reason, the current ECCO-EFCCA patient guidelines strongly recommend regular psychiatric evaluation as a necessary part of patients' standard follow-up and put particular emphasis on treating anxiety and depressive symptoms with the use of appropriate pharmacological or psychosocial interventions. However, relevant literature is relatively sparse, lacking wide-scale randomized trials focusing on the efficacy of antidepressants and psychotherapy not only on alleviating patients' psychological distress but also on improving IBD clinical and laboratory severity indices. More specifically, a recent systematic review identified only one randomized clinical trial on the effect of antidepressants in IBD patients. In a similar vein, there is a limited number of randomized clinical trials focusing on the effect of brief psychotherapeutic interventions on patients' psychological burden, QoL and disease progression.

The importance of different immunoregulatory pathways mediated by several immunological cells subtypes and cytokines in the regulation of IBD has been demonstrated the last years. Cytokines have been directly implicated in the pathogenesis of IBD in genetic and immunological studies, and they establish a crucial role in controlling intestinal inflammation and the associated clinical symptoms of IBD. Despite the fundamental role of cytokines in controlling mucosal inflammation in IBD, to our knowledge, inflammation indices have never been evaluated as study end-points in investigations focusing on the role of psychotherapy on patients' QoL.

Research hypotheses Our primary research hypothesis is that brief psychotherapeutic intervention will reduce IBD patients' gastrointestinal symptoms and psychological distress and improve their sexual functioning and QoL. A secondary hypothesis is that the observed improvement in psychosocial functioning will be accompanied by alterations in inflammation and disease activity indices.

Research aim In this context, the aim of the current prospective randomized controlled study will be the measurement of the effects of brief group cognitive behavioral psychotherapy on gastrointestinal symptom severity, psychological distress, sexual functioning, QoL and inflammation and disease activity indices in IBD patients. An additional aim will be the detection of psychological and biomedical parameters which are associated with these effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients suffering from Crohn's disease or ulcerative colitis according to the ECCO-EFCCA Patient Guidelines, in both statuses "currently experiencing a flare/relapse" or "not currently experiencing a flare/relapse (in remission)"

Exclusion Criteria:

* major psychopathology
* severe cognitive or neurological deficits
* cancer
* other severe chronic diseases or disabilities
* lack of fluency in the Greek language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Health Survey 36 Short Form (SF36) | 18 months
  The SF36 is a self-report, generic quality of life instrument, which includes eight multi-item scales (36 items) that evaluate the extent to which an individual's health limits his or her physical, emotional, and social well-being. The SF-36 covers eight domains of HRQOL, namely physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems, and mental health. Scores on each subscale range from 0 to 100, with higher scores indicating a better quality of life. Sub-scales scores are calculated according to an algorithm described in the SF36 manual.
Hospital Anxiety and Depression Scale (HADS) | 18 months
  This is a widely used psychometric tool, comprised of 14 items, 7 items for anxiety and 7 items for depression. Each subscale is scored from 0-21. Higher scores indicate greater severity of depressive and anxious symptoms
Female Sexual Functioning Index (FSFI) | 18 months
  The FSFI is a 19-item questionnaire which measures 6 domains, namely sexual desire, arousal (both subjective and physiologic), lubrication, orgasm, satisfaction and pain. The 6 domain scores are summed to produce a full-scale score. For all FSFI domains, higher values indicate a better level of functioning
International Index of Erectile Function(IIEF) | 18 months
  This is a 15-item, validated questionnaire which has proven extremely useful in the clinical assessment of erectile dysfunction and has been widely used in clinical trials to evaluate treatment outcomes. Each question can be awarded a score between 0 and 5 and the questionnaire as a whole addresses the main four domains of male sexual functioning (erectile functioning, orgasmic functioning, sexual desire and intercourse satisfaction) along with a fifth component which encompasses the concept of overall sexual satisfaction

SECONDARY OUTCOMES:
Crohn's disease activity index | 6 months
  This is an index measuring the severity of Crohn's Disease. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease, and values above 450 are seen with extremely severe disease.
Truelove and Witts' severity index | 6 months
  This is an index which classifies adult patients with ulcerative colitis into 3 categories (mild, moderate, severe) based on clinical signs and laboratory values.
Feacal calprotectin | 6 months
  Faecal calprotectin is a biochemical measurement of the protein calprotectin in the stool. Elevated faecal calprotectin indicates the migration of neutrophils to the intestinal mucosa, which occurs during intestinal inflammation, including inflammation caused by inflammatory bowel disease.
Serum cytokines levels | 6 months
  Cytokines are chemical substances involved in inflammatory processes. Their levels are altered in chronic inflammation such as in ulcerative colitis and Crohn's Disease

CONTACTS AND LOCATIONS:
Overall Officials: Christos Triantos, PhD, Principal Investigator — University of Patras, Medical School
Locations (1):
- Department of Gastroenterology, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrne G, Rosenfeld G, Leung Y, Qian H, Raudzus J, Nunez C, Bressler B. Prevalence of Anxiety and Depression in Patients with Inflammatory Bowel Disease. Can J Gastroenterol Hepatol. 2017;2017:6496727. doi: 10.1155/2017/6496727. Epub 2017 Oct 18. PMID 29181373
- [Background] Limsrivilai J, Stidham RW, Govani SM, Waljee AK, Huang W, Higgins PD. Factors That Predict High Health Care Utilization and Costs for Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2017 Mar;15(3):385-392.e2. doi: 10.1016/j.cgh.2016.09.012. Epub 2016 Sep 17. PMID 27645518
- [Background] Macer BJ, Prady SL, Mikocka-Walus A. Antidepressants in Inflammatory Bowel Disease: A Systematic Review. Inflamm Bowel Dis. 2017 Apr;23(4):534-550. doi: 10.1097/MIB.0000000000001059. PMID 28267046
- [Background] Schoultz M, Atherton I, Watson A. Mindfulness-based cognitive therapy for inflammatory bowel disease patients: findings from an exploratory pilot randomised controlled trial. Trials. 2015 Aug 25;16:379. doi: 10.1186/s13063-015-0909-5. PMID 26303912
- [Background] McCombie A, Gearry R, Andrews J, Mulder R, Mikocka-Walus A. Does Computerized Cognitive Behavioral Therapy Help People with Inflammatory Bowel Disease? A Randomized Controlled Trial. Inflamm Bowel Dis. 2016 Jan;22(1):171-81. doi: 10.1097/MIB.0000000000000567. PMID 26360545
- [Background] Mikocka-Walus A, Bampton P, Hetzel D, Hughes P, Esterman A, Andrews JM. Cognitive-Behavioural Therapy for Inflammatory Bowel Disease: 24-Month Data from a Randomised Controlled Trial. Int J Behav Med. 2017 Feb;24(1):127-135. doi: 10.1007/s12529-016-9580-9. PMID 27432441
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Kalogeropoulou M, Karaivazoglou K, Konstantopoulou G, Vinni E, Sotiropoulos C, Tourkochristou E, Aggeletopoulou I, Lourida T, Labropoulou E, Diamantopoulou G, Mouzaki A, Assimakopoulos K, Gourzis P, Thomopoulos K, Theocharis G, Triantos C. The Impact of Group Cognitive Behavioral Psychotherapy on Disease Severity and Psychosocial Functioning in Patients With Inflammatory Bowel Disease: A Randomized Controlled Study. J Crohns Colitis. 2025 Mar 5;19(3):jjae144. doi: 10.1093/ecco-jcc/jjae144. PMID 39316575